CLINICAL TRIAL: NCT04556448
Title: A Randomized Controlled Trial Comparing the Effectiveness of Invisalign and Traditional Orthodontic Treatments
Brief Title: RCT Comparing Invisalign and Traditional Orthodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Peter H. Buschang, Professor, Orthodontics, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-21_COD_Ortho1
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Malocclusion, Angle Class II
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Orthodontic Appliances, Removable

STUDY DESIGN:
Intervention Model Description: Randomized RCT
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aligners (Experimental): Invisalign treatment
  Interventions: Other: Aligners
- Traditional braces (Active Comparator): Clear braces
  Interventions: Other: Clear braces

INTERVENTIONS:
Other: Aligners — Clear aligners
  Other Names: Invisalign
  Arms: Aligners
Other: Clear braces — Clear braces
  Arms: Traditional braces

SUMMARY:
Comparison of orthodontic patients treated with aligners and traditional (clear braces)

DETAILED DESCRIPTION:
Patients were selected based on being adults and having mild Class I malocclusion. They were randomly allocated into either the aligner group and the traditiona (clear braces group).. The aligner group was treated with invisalign, with up to two adjustments at the end of treatment. The traditional group had clear braces placed on their teeth. The outcome variables including the following: 1) pain and discomfort related to treatment, 2) posttreatment occlusal status, and 3) postretention occlusal status.

ELIGIBILITY:
Inclusion Criteria:

1. Class I molar and canine relationships
2. Non-extraction treatments
3. Mandibular crowding of 4 mm or less
4. No missing tooth (from second to second molar)

Exclusion Criteria:

1. Anterior or posterior crossbites
2. Anterior or lateral open bites
3. Maxillary overjet exceeding 3mm
4. Impacted tooth

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Occlusal changes | up to 6 months
  Differences in occlusion between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Peter Buschang, PhD, Principal Investigator — TAMU Health Science Center
Locations (1):
- Texas A&M Baylor College of Dentisry, Dallas, Texas, United States